CLINICAL TRIAL: NCT07276711
Title: Controlled Arterial Protection to Ultimately Remove Embolic Material
Brief Title: CAPTURE-2: Controlled Arterial Protection to Ultimately Remove Embolic Material
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EmStop Inc (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS-CL-5100
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Aortic Valve Stenosis; Aortic Stenosis; Aortic Valve Disease
Keywords: Transcatheter aortic valve replacement (TAVR); Cerebral embolic protection device; Stroke; Cerebrovascular accident; Neuroprotection; Aortic valve disease; Aortic valve stenosis; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be blinded to their treatment assignment to minimize expectation and reporting bias. Procedural teams will be unblinded due to the nature of device deployment; the device is temporary and not intended for implantation. Every effort will be made to have follow-up personnel remain blinded, with those conducting the neurological assessments being most critical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- EmStop System (Experimental)
  Interventions: Device: EmStop Embolic Protection System
- Boston Scientific Sentinel device (Active Comparator)
  Interventions: Device: Boston Scientific Sentinel

INTERVENTIONS:
Device: EmStop Embolic Protection System — EmStop Embolic Protection System used during TAVR procedure
  Arms: EmStop System
Device: Boston Scientific Sentinel — Sentinel device used during TAVR procedure
  Arms: Boston Scientific Sentinel device

SUMMARY:
The objective of this study is to demonstrate safety and efficacy of the EmStop Embolic Protection System when used as indicated to capture and remove thrombus/debris during self-expanding transcatheter aortic valve replacement (TAVR) procedures.

DETAILED DESCRIPTION:
This is a prospective, single-blind, multi-center, randomized study conducted in up to 25 U.S. investigational sites. Subjects with severe aortic valve stenosis (AS) will be randomized 2:1 to the EmStop Embolic Protection System (study device) versus the Sentinel device (control group) and followed to 30 days post TAVR procedure.

ELIGIBILITY:
Clinical Inclusion Criteria

1. Age ≥ 22 years at the time of consent
2. Meets FDA-approved indications for elective transfemoral self-expanding transcatheter aortic valve replacement (TAVR) procedure on a native or non-native (valve-in-valve) aortic valve. Note: Due to Neurologist availability and importance of capturing the neurological assessments, procedures must be performed Monday-Thursday.
3. Left ventricular ejection fraction ≥ 30% as confirmed by echocardiogram
4. Willing and able to provide written informed consent and written HIPAA authorization prior to initiation of study procedures
5. Willing and able to comply with the protocol-specified procedures and assessments

Imaging Inclusion Criteria

1. Echocardiogram including left ventricular ejection fraction ≥ 30% within 6 months (180 days) prior to the index procedure and prior to randomization to confirm adequate cardiac function.
2. Subjects must undergo a computed tomography angiography (CTA) scan within 6 months (180 days) prior to the index procedure and prior to randomization to confirm anatomic compatibility with the study device and the control device. Subjects must meet the following anatomical inclusion criteria:

EmStop Angiographic (CTA) Inclusion Criteria 1. Subject anatomy is compatible with correct device positioning with:

* Ascending aorta length ≥8 cm
* Femoral and iliac artery minimal lumen diameter of ≥ 8.0 mm
* Ascending aorta/aortic arch diameter is ≥25 or ≤40 mm.
* Ascending aorta or aortic arch exhibits ≤ Grade 1 atheromatous disease and limited wall calcification

Sentinel Angiographic (CTA) Inclusion Criteria

1. Subject anatomy, excluding bovine arch anatomy, is compatible with correct device positioning with:

* Artery diameter is 9-15 mm for the brachiocephalic artery and 6.5-10 mm in the left common carotid artery
* Arterial stenosis <70% in either the left common carotid artery or the brachiocephalic artery
* Brachiocephalic or left carotid artery without significant stenosis, ectasia, dissection, or aneurysm at the aortic ostium or within 3 cm of the aortic ostium
* Adequate blood flow to the right upper extremity
* Access vessels without excessive tortuosity

Exclusion Criteria:

1. Requires use of a balloon-expandable transcatheter aortic valve for the index procedure
2. Documented history of stroke or transient ischemic attack (TIA) within the prior 6 months, or any prior stroke with a permanent major disability or deficit (National Institute of Health Stroke Scale [NIHSS] >1 at baseline)
3. Left ventricular ejection fraction <30%, cardiogenic shock, or hypotension requiring inotropes or mechanical circulatory support, within 3 months prior to index procedure
4. Acute myocardial infarction (MI) within 30 days of the planned index procedure
5. Planned to undergo any other open cardiac surgical or left heart interventional procedure (e.g., concurrent coronary revascularization) during the TAVR procedure or within 30 days prior to the TAVR procedure. The need for a postoperative pacemaker implant after TAVR is not exclusionary.
6. Renal failure, defined as estimated glomerular filtration rate (eGFR) <30 mL/min
7. Hypercoagulable state that cannot be corrected by additional periprocedural heparin
8. History of intolerance, allergic reaction, or contraindication to any of the study medications, including heparin, aspirin, clopidogrel, or a sensitivity to contrast media or anesthesia that cannot be adequately pre-treated
9. Undergoing therapeutic thrombolysis
10. History of bleeding diathesis or major coagulopathy
11. Hepatic failure (Child-Pugh class C)
12. Active endocarditis or ongoing systemic infection, defined as fever (>38°C) and/or WBC >15,000 IU
13. Known allergy to any materials used in the EmStop system (e.g., nitinol)
14. Currently participating in another drug or device clinical study
15. Known or suspected to be pregnant, or is lactating; women of child bearing age must have a negative serum or urine pregnancy test within 48 hours prior to the index study procedure
16. Vulnerable subject populations (e.g., incarcerated or cognitively challenged adults)
17. Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Non-Inferiority | Non-inferiority of 30-day EmStop device MACCE patient incidence rate compared to the Sentinel device patient incidence rate
  Primary combined safety and efficacy endpoint is the rate of major adverse cardiac and cerebrovascular events (MACCE) at 30-days

SECONDARY OUTCOMES:
Non-Inferiority | 30 days
  Hypothesis-driven secondary efficacy endpoint is the composite rate through 30-days post-procedure of NeuroARC defined ischemic embolic stroke, VARC-3 defined AKI, and systemic embolization
Debris Capture | 30 days
  Hypothesis-driven secondary efficacy endpoint is the total debris capture, defined as the number of captured particles of at least ≥ 150micron

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Chetcuti, MD, Principal Investigator — University of Michigan Health

IPD SHARING:
Plan to Share IPD: No